CLINICAL TRIAL: NCT07067333
Title: Elastic Intramedullary Nails Versus Plate Fixation in Treatment of Diaphyseal Femoral Fracture in Adolescent
Brief Title: Fixation of Shaft Femure Fracrture by Ender Versus Plate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Hashem Ahmed, lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-5-4MS
Record Dates: First submitted 2025-06-23; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Shaft Femure Fracture in Adolescents
MeSH Terms: interventions — Fracture Fixation, Intramedullary; Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A for intramadullary nail (Active Comparator): fixation of the femure in group A by intramedullary nails
  Interventions: Device: intramedullary nails for group A
- group B for plating (Active Comparator): fixation of the shaft femure fracture in group B by plates
  Interventions: Device: plate for group B

INTERVENTIONS:
Device: intramedullary nails for group A — fixation of the shaft femure fracture in this group by intramedullary nails
  Arms: group A for intramadullary nail
Device: plate for group B — fixation of the shaft femure fracture in the group b by plates
  Arms: group B for plating

SUMMARY:
The aim of this study is to compare the

* functional outcomes, fracture healing time, rate of complications, and long-term growth outcomes between intramedullary nail and plating in adolescent.
* Assess radiographic outcomes (e.g., alignment, limb length discrepancy, and growth plate disturbance).
* Evaluate complications such as infection, nonunion, malunion, refractures, and need for reoperation (e.g., hardware removal).

DETAILED DESCRIPTION:
Elastic Nails (EN) are flexible intramedullary devices, usually made of titanium or stainless steel, that allow for dynamic stabilization. They are typically used for fractures in children and adolescents. The intramedullary nails offer the advantage of minimally invasive insertion, less disruption of the periosteum, and potential for less disruption of the growth plate.The nails bend and allow for some motion at the fracture site, which promotes healing through the formation of callus.

Plate fixation typically involves a compression or neutralization plate, usually a dynamic compression plate (DCP) or a locking plate. This method provides rigid stabilization but often requires more extensive dissection and can interfere with growth if the plate is applied too close to the physis (growth plate).While plating can be very effective in providing stability, there is a higher risk of complications such as hardware-related issues (e.g., plate prominence, need for removal) and potential growth disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-16 years (skeletally immature, based on radiographic evidence of growth plates).
* Diagnosis: Closed or open (Grade I) diaphyseal femoral fractures.
* Fracture type: Simple transverse, short oblique, or spiral fractures (classified by the AO/OTA system or by the Müller classification).

Exclusion Criteria:

* • Fractures with significant comminution or open fractures (Grade II or III).

  * Pathological fractures (e.g., secondary to bone disease).
  * Severe systemic conditions that may affect bone healing or postoperative recovery (e.g., metabolic bone diseases).
  * Patients with previous ipsilateral femur fractures or those requiring re-operation for non-union or malunion.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Fracture Femure fixation by intramedullary nails versus plates | 6 months
  limb length discrepancy by planning X rays.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No